CLINICAL TRIAL: NCT02445885
Title: Late Reperfusion With Percutaneous Coronary Intervention in Patients With ST-segment Elevation Myocardial Infarction
Acronym: LATE-MI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Engstrom (Other)
Responsible Party: Sponsor-Investigator, Thomas Engstrom, Chief Consultant, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LATE-MI
Record Dates: First submitted 2015-05-08; First posted 2015-05-15 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Heart Disease; ST-segment Elevation Myocardial Infarction
Keywords: Myocardial infarction; Late presenters; Primary percutaneous coronary intervention; Reperfusion; Angioplasty; Duration of ischemia; Cardiovascular magnetic resonance imaging
MeSH Terms: conditions — Myocardial Ischemia; ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acute PCI (Experimental): Acute re-opening of the occluded coronary artery including premedication as for primary PCI within 12 hours
  Interventions: Procedure: PCI
- Subacute PCI (Active Comparator): Standard subacute re-opening of the occluded coronary artery including premedication as for subacute PCI within 72 hours
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — Guideline directed Percutaneous Coronary Intervention

SUMMARY:
Although recommended therapy for patients with ST-segment elevation myocardial infarction is primary PCI, it remains unestablished whether patients with a symptom duration of more 12 hours benefit from acute revascularisation.

This study aims to investigate whether acute intervention is superior to subacute intervention in these patients.

DETAILED DESCRIPTION:
The recommended therapy for patients with ST-segment elevation myocardial infarction (STEMI) is to restore normal coronary blood flow with timely reperfusion by percutaneous coronary intervention (PCI), and thereby minimize the extent of cell death and preserving cardiac function. The duration of ischemia and timely PCI are major determinants for the size of the myocardial infarction and prognosis. Thus, acute PCI should be performed within 12 hours after symptom onset. The effect of PCI and timing of PCI are, however, much more uncertain for late presenters who contact the health service > 12 hours from symptom. Thus, it is still unknown whether late presenters should be treated with acute PCI or medical treatment with delayed PCI (24-72 h after first medical contact).

The study investigates the effect on final salvage index evaluated by magnetic resonance imaging of acute PCI of late presenters.

The overall objective of the study is to investigate whether late presenters may benefit from acute PCI, and thus whether to extend the currently recommended time limit of 12 hours for acute PCI in patients with STEMI.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Patients more than 18 years of age.
* STEMI > 12 hours and < 36 hours.
* Clinical stable, i.e. no on going angina, hemodynamically stable (systolic BP > 90) and Killip class < 3.

Exclusion Criteria:

* Clinical instability which requires an acute invasive strategy.
* Left main occlusion or multivessel disease which requires CABG.
* Previous Q-wave infarction in the current infarct related artery.
* Left Bundle Branch Block (LBBB).
* Severe renal insufficiency.
* Pacemaker
* Chronic atrial fibrillation.
* Previous Coronary Artery Bypass Surgery (CABG).
* Pregnancy.
* Other severe illness with life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-05; Primary Completion 2024-03-01 (Estimated); Study Completion 2039-03-01 (Estimated)

PRIMARY OUTCOMES:
Acute salvage index evaluated by MRI | 1-2 days
  MRI within 48 timer after index admission will be used to measure are at risk (AAR, T2-weighted) and acute infarct size (IZ). Acute salvage index is (AAR-IZ)/AAR

SECONDARY OUTCOMES:
Final infarct size | 3 months
  Please see above
Final myocardial salvage index | 1-2 days
  As for primary endpoint but IZ is measured within the index admission
Acute infarct size | 1-2 days
Microvascular obstruction (MVO) | 1-2 days
Left Ventricular Ejection Fraction (LVEF) | 1-2 days and 3 months
  Measured by MRI

OTHER OUTCOMES:
Left Ventricular (LV) volumes | 1-2 days and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nepper-Christensen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Background] Terkelsen CJ, Sorensen JT, Maeng M, Jensen LO, Tilsted HH, Trautner S, Vach W, Johnsen SP, Thuesen L, Lassen JF. System delay and mortality among patients with STEMI treated with primary percutaneous coronary intervention. JAMA. 2010 Aug 18;304(7):763-71. doi: 10.1001/jama.2010.1139. PMID 20716739
- [Background] Carlsson M, Ubachs JF, Hedstrom E, Heiberg E, Jovinge S, Arheden H. Myocardium at risk after acute infarction in humans on cardiac magnetic resonance: quantitative assessment during follow-up and validation with single-photon emission computed tomography. JACC Cardiovasc Imaging. 2009 May;2(5):569-76. doi: 10.1016/j.jcmg.2008.11.018. PMID 19442942
- [Result] Busk M, Kaltoft A, Nielsen SS, Bottcher M, Rehling M, Thuesen L, Botker HE, Lassen JF, Christiansen EH, Krusell LR, Andersen HR, Nielsen TT, Kristensen SD. Infarct size and myocardial salvage after primary angioplasty in patients presenting with symptoms for <12 h vs. 12-72 h. Eur Heart J. 2009 Jun;30(11):1322-30. doi: 10.1093/eurheartj/ehp113. Epub 2009 Apr 8. PMID 19357105
- [Result] Schomig A, Mehilli J, Antoniucci D, Ndrepepa G, Markwardt C, Di Pede F, Nekolla SG, Schlotterbeck K, Schuhlen H, Pache J, Seyfarth M, Martinoff S, Benzer W, Schmitt C, Dirschinger J, Schwaiger M, Kastrati A; Beyond 12 hours Reperfusion AlternatiVe Evaluation (BRAVE-2) Trial Investigators. Mechanical reperfusion in patients with acute myocardial infarction presenting more than 12 hours from symptom onset: a randomized controlled trial. JAMA. 2005 Jun 15;293(23):2865-72. doi: 10.1001/jama.293.23.2865. PMID 15956631